CLINICAL TRIAL: NCT05921318
Title: The Safety and Efficiency of Beijing Protocol in Malignant Hematologic Disease Patients Receiving More Than 5/10 HLA-mismatched Allo-HSCT
Brief Title: Beijing Protocol in Patients Receiving More Than 5/10 HLA-mismatched Allo-HSCT
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, director, hematology department,Peking University People's Hospital, Peking University People's Hospital
Other Study IDs: Highly HLA mismatched HSCT
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Hematologic Malignancy; Stem Cell Transplant Complications
Keywords: allogenetic hematopoietic stem cell transplant; HLA locus; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- more than 5/10 HLA-mismatched allo-HSCT: more than 5/10 HLA-mismatched allo-HSCT
  Interventions: Combination Product: Beijing protocol

INTERVENTIONS:
Combination Product: Beijing protocol — For patients <55 years and HCT-CI≤ 3：Ara-C(4g/m2/day,-9 days),Bu(9.6mg/kg,-8 days to -6 days),Cy(1,800mg/m2/day,-5 days to -4 days),semustine(250mg/m2,-3 days),ATG(7.5-10 mg/kg,-5 to -2 days)
  For patients ≥ 55 years or HCI-CI>3：Ara-C(2g/m2/day,-10 days to -9 days),Bu(9.6mg/kg,-8 days to -6 days),Flu(30mg/m2/day,-6 days to -2 days),Cy(1,000mg/m2/day,-5 days to -4 days),semustine(250mg/m2,-3 days),ATG(7.5-10 mg/kg,-5 to -2 days).

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of Beijing protocol in malignant haematologic disease patients receiving more than 5/10 HLA-mismatched allo-HSCT.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is a potentially curative procedure for patients with hematological malignancies.Donor-recipient human leukocyte antigen (HLA) compatibility plays a key role in successful allo-HSCT as HLA-matching has a direct impact on the risk of GvHD, non-relapse mortality (NRM), and survival. Suitable, matched or haploidentical donors are not always available or accessible, even in the era of the international registries.Therefore, there is a need for new strategies that could negate the barrier of HLA-mismatching, allowing allo-HSCT from traditionally prohibitive highly mismatched donors.The aim of the study is to evaluate the efficacy and safety of Beijing protocol in malignant haematologic disease patients receiving more than 5/10 HLA-mismatched allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* hematologic malignancy patients
* patients eligible for the transplantation of allogeneic hematopoietic stem cells;
* patients unavailable with HLA matched donor or related haploidentical donor
* voluntary participation in this study and signing the informed consent form.

Exclusion Criteria:

* Patients with the severe infections;
* Pregnant or lactating women
* Patients who are not eligible for hematopoietic stem cell transplantation;
* Patients who are enrolled in other clinical trials within 1 month;
* Patients who may not be able to complete the study for other reasons, or may be considered by the investigator not suitable to participate in the study;
* Patients unable to properly understand or refusing to accept the informed consent form.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with hematologic malignancy，unavailable with HLA matched donor or related haploidentical donor
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
1-year LFS | Participants will be followed for an expected average of 1 years
  defined as disease relapse, disease progression or death (whichever occurs first) within 1 year from the day the patient receives transplantation.

SECONDARY OUTCOMES:
1-year OS | Participants will be followed for an expected average of 1 years
  defined as survival rate within 1 year from the day the patient receives transplantation, calculated based on death from any cause.
1-year TRM | Participants will be followed for an expected average of 1 years
  defined as death from any cause other than disease relapse within 1 year from the day the patient receives transplantation.

OTHER OUTCOMES:
Adverse event | Participants will be followed for an expected average of 1 years
  The incidence rate of acute GVHD, chronic GVHD, CMV activation, EBV activation after transplantation
Engraftment rate | Participants will be followed for an expected average of 1 years
  The success rate of engraftment after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Prof., Principal Investigator — Peking University People's Hospital
Locations (1):
- Deparment of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided